CLINICAL TRIAL: NCT04373668
Title: Reducing Hypnotic Drug Use and Improving Night-time Care for People Living With Dementia in Care Homes (NightCAP): A Randomised Factorial Trial
Brief Title: NightCAP: Reducing Hypnotic Drug Use and Improving Night-time Care
Acronym: NightCAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Exeter (Other)
Collaborators: King's College London (Other); University of East Anglia (Other); Aston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1920/13
Record Dates: First submitted 2020-04-28; First posted 2020-05-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Dementia
Keywords: Dementia; Care Homes; Hypnotic Medication; Night Time Care; Behavioural symptoms; Cost effectiveness
MeSH Terms: conditions — Dementia; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, optimised usual care (No Intervention): Treatment delivered as usual in the care home
- Hypnotic Drug Review, Structured Sleep Hygiene and NightCAP (Experimental): Care homes to receive all three interventions: Hypnotic Drug Review, Structured Sleep Hygiene and NightCAP interventions
  Interventions: Behavioral: Hypnotic Medication Review; Behavioral: Structured Sleep Hygiene; Behavioral: Night Time Care Activities Programme

INTERVENTIONS:
Behavioral: Hypnotic Medication Review — A training programme focused providing guidance on the review and withdrawal process of hypnotic drugs.
  Arms: Hypnotic Drug Review, Structured Sleep Hygiene and NightCAP
Behavioral: Structured Sleep Hygiene — Training module on the principle of good sleep hygiene
  Arms: Hypnotic Drug Review, Structured Sleep Hygiene and NightCAP
Behavioral: Night Time Care Activities Programme — Training and support package to assist in the development of a personalised night time care plan and support the implementation and dissemination of information within the care home environment
  Arms: Hypnotic Drug Review, Structured Sleep Hygiene and NightCAP

SUMMARY:
Dementia is a devastating condition characterised by progressive loss of cognition leading to loss of independence and eventually death. One major unmet need, which remains a critical challenge for care provision, is the management of night-time care and sleep-related symptoms in people with dementia living in care homes. The causes and impacts of sleep disturbances in people with dementia in care homes are complex and multi-faceted, indicating the need of a whole-systems approach to the issue. It will require a tailored, person-centred approach which accounts for the environmental, personal and clinical factors contributing to the symptoms.

The aim of this study is to evaluate the NightCAP intervention to improve treatment of sleep disturbance in people with dementia in care homes, with the goal of reducing sleep disturbance behaviour and reducing the use of hypnotic drugs. This will provide robust evidence to support guidance on night time care and improving hypnotic drug prescribing, both of which are major unmet needs in the care of people with dementia.

DETAILED DESCRIPTION:
The main objective of this current study is to explore the effectiveness of specific benefits of key components of the Night Time Care Activities Programme- NightCAP. Particularly elements of sleep hygiene and personalised night-time care planning. There may also be additional benefit in combining NightCAP elements with pharmacological review protocol to enable management of all major contributing factors in sleep disturbance.

This cluster-randomised trial will be delivered in 24 UK care homes. Participants will be individuals living with dementia and experiencing sleep disturbance, as well as staff who care for them. Homes will be randomly allocated to one of two arms: optimised usual care or the intervention arm. All homes will receive an optimised person-centred care module. The NightCAP intervention programme consists of three key elements: (i) personalised night-time care planning (supported staff training and implementation); (ii) structured sleep hygiene (staff training); and (iii) hypnotic drug review protocol (GP fact sheet and staff training). The primary outcome will be sleep disturbance at the end of the intervention. Secondary outcomes will be hypnotic drug use, quality of life, resident falls, job satisfaction, burden and coping in care staff, and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Care homes (inclusive of residential and nursing) that have failed to meet more than 1 of the 5 CQC care home quality standards check
* Care homes who have at least 12 eligible care home resident participants
* Care homes with a minimum of two residents who are eligible to participate in the study taking hypnotic medication
* Resident participants will have an established or probable diagnosis of dementia
* Residents will have experienced an episode/occurrence of sleep disturbance behaviour in the past four weeks/two weeks (as reported by care staff)
* Care home member of staff whose duties include providing care to individuals with dementia
* Care home care staff are required to have an adequate level of English language to complete all required assessment outcomes
* Care home care staff participants who will remain in work without plans for extended leave over the study period

Exclusion Criteria:

* Care homes receiving special support from the local authority
* Agency care staff
* Care staff will be able to withdraw from the study at any time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Disturbance Inventory SDI | From baseline and immediately after intervention
  Sleep disturbance behaviour as measured by the Sleep Disturbance Inventory SDI

SECONDARY OUTCOMES:
Change of Hypnotic Drug Use | From baseline, immediately after intervention and at four months follow-up
  Hypnotic drug use assessed from the care home Medication Administration Record
Dementia Quality of Life | From baseline, immediately after intervention and at four months follow-up
  Quality of life assessed using DEMQOL-Caregiver. Consisting of 32 questions the DEMQOL-Caregiver is an interviewer administered measure, with higher scores indicating better quality of life.
Neuropsychiatric Inventory- Nursing Home (NPI-NH) | From baseline, immediately after intervention and at four months follow-up
  The NPI is a validated structured interview assessment with the informant (care staff), that assesses behavioural disturbances in patients with dementia. This 12-item version consists of 10 behavioural and two neurovegetative areas. It provides both a total score as well as scores for a number of sub-scales (e.g. delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, disinhibition, elation/euphoria, apathy/indifference, irritability/lability, aberrant motor activity, sleep, and appetite/eating disorders). The frequency, severity and caregiver distress for each domain are measured. The total possible maximum score is 144. A higher score reflects increased frequency and severity of the disturbances. This specific version is developed for use in care homes, with adapted questions in the standardised interview and the caregiver distress assessment adapted to occupation disruptiveness.
Cohen-Mansfield Agitation Inventory (CMAI) | From baseline, immediately after intervention and at four months follow-up
  The CMAI is a caregivers' rating questionnaire to specify agitated behaviour (Cohen-Mansfield et al, 1980). The CMAI consist of 29 items related to agitated behaviour, each of which is rated on a 7- point scale of frequency, from 1= never to 7= several times an hour. The rating is based on a face-to-face interview with a caregiver.
Global Deterioration Scale (GDS) | From baseline, immediately after intervention and at four months follow-up
  The GDS is a staging scale indicating deterioration in dementia. The scale details clinical descriptions of seven major distinguishable stages, ranging from normal cognition to severe dementia. Stages 1-3 are the pre dementia stages/ Stages 4-7 reflect the stages of dementia.
Client Service Receipt Inventory (CSRI) | From baseline, immediately after intervention and at four months follow-up
  The CSRI is used to estimate the cost of service packages for each participant in the study. Information is collected on the current living arrangements, use of hospital, community-based and day services. The data collected through the CSRI can be used to calculate service costs and total costs of care.
Functional Assessment Staging (FAST) | From baseline, immediately after intervention and at four months follow-up
  FAST is a proxy-rated instrument validated for use in people with dementia. It ascertains the severity of dementia in seven stages of functioning.
EQ5D-5L | From baseline, immediately after intervention and at four months follow-up
  The EQ5D-5L is a measure of Health Related Quality of Life. The EQ5D-5L consist of the EQ5D descriptive system and the EQ visual analogue scale (EQ VAS).
Abbey Pain Scale | From baseline, immediately after intervention and at four months follow-up
  The Abbey Scale is an observation brief indicator of pain for people with end-stage dementia. The scale is rated on six non verbal indicators of pain where 0 is none and 3 is severe
Approached to Dementia Questionnaire (ADQ) | From baseline, immediately after intervention and at four months follow-up
  The ADQ is a 19-item instrument. Responses are indicated using a 5-point Likert scale. Higher values represent a better outcome (range from 19-96). The ADQ includes two subscales: person-centredness and hopefulness.
Patient Health Questionnaire 9 (PHQ-9) | From baseline, immediately after intervention and at four months follow-up
  A measure of carer mental health and behaviour consisting of 9 questions

CONTACTS AND LOCATIONS:
Overall Officials: Anne Corbett, Study Chair — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No